CLINICAL TRIAL: NCT06698094
Title: Impact of a Sustainable Lifestyle on Dietary Quality, CO2e Emissions and Physical Activity in Office Workers: a Study Protocol for a Cluster Randomized Controlled Trial (SOFIA Project)
Brief Title: Sustainable Office Intervention, Impact of a Sustainable Lifestyle on Diet, Physical Activity and Carbon Footprint
Acronym: SOFIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mälardalen University (Other)
Collaborators: Swedish Environmental Research Institute (IVL) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-2020/0244
Record Dates: First submitted 2024-08-08; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Healthy Lifestyle; Healthy Diet
Keywords: Sustainability; Physical activity; Active transportation; Dietary fiber; Organic food
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A two-arm parallel cluster randomized trail
Who Masked: Participant
Masking Description: Participants will be recruited without knowledge of differences between the two arms, and cluster randomized based on there working space (office) with allocation concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy lifestyle group (HL) (Active Comparator): The control group will receive advice about a conventional healthy diet according to the Nordic Nutrition Recommendations (NNR 2014) and international physical activity recommendations from WHO. The participants will get information about the recommended distribution of energy from macronutrients i.e. energy coming from fat, protein, and carbohydrates, as well as general recommendations about the "plate model", i.e. the combination of food on the plate to adhere to the recommended nutrient intake. Additionally, they will receive instructions to increase physical activity to reach 150 to 300 minutes of moderate aerobic activity per week or the equivalent vigorous activity.
  Interventions: Behavioral: Healthy lifestyle
- Sustainable lifestyle group (SL) (Experimental): The sustainable lifestyle group will receive instructions to increase the consumption of healthy organic plant-based foods that is carbon or environmentally friendly (i.e. fruits, vegetables, legumes, multigrain cereals, or labeled foods) and decrease consumption of beef and dairy products. We expect that the reduction of diet-related CO2e will be 50% as compared to the baseline, while the intake of nutrients such as fiber, vitamin C, and folate will increase. Additionally, they will receive instructions to increase active and emission-free transportation, i.e. walking and biking to and from work and meetings.
  Interventions: Behavioral: Sustainable lifestyle

INTERVENTIONS:
Behavioral: Sustainable lifestyle — To encourage and nudge a sustainable lifestyle in an office context in order to improve public health and combat climate change.
  Arms: Sustainable lifestyle group (SL)
Behavioral: Healthy lifestyle — To encourage and nudge a healthy lifestyle in an office context, the participants in this arm will function as a control group receiving general recommendations based on NNR 2014 nutritional recommendations and WHO physical activity recommendations.
  Arms: Healthy lifestyle group (HL)

SUMMARY:
The main goal of the study, Sustainable Office Intervention (SOFIA), is to promote and ease the adoption of a sustainable lifestyle within an office environment, with the dual goals of enhancing public health and mitigating the adverse effects of climate change. Specifically, the study aims to assess the effectiveness of promoting sustainable lifestyle choices in the office workplace compared to promoting a conventional healthy lifestyle in regards to diet and physical activity.

DETAILED DESCRIPTION:
The participants will be recruited at companies in the Swedish office sector, and after recruitment and baseline assessment, the participants will be randomly assigned to one of two groups Healthy Lifestyle (HL) or Sustainable Lifestyle (SL).

All participants will complete web-based questionnaires including background information about weight, height, diet, physical activity, smoking, education and other relevant background variables at the beginning of the study as well as at the end of the study. Participants will attend separate group-based workshops 6 times during the 8-week intervention period held by trained personnel. During these workshops, participants will be guided by education, food provision, and assistance to identify facilitators and barriers to a healthy or sustainable lifestyle. In addition, adherence to a healthy or sustainable lifestyle will be reinforced using a behavioral support package provided through a digital platform during the intervention period.

We will compare baseline, midpoint, and final (i.e. week 0, 4 and 8) nutrient intake, CO2e, and the dietary sustainability score for the two diets with an ANOVA model. We assume a dropout rate of 10-15% after baseline assessment (based on our previous pilot study from the fall of 2017) Climate Friendly and Ecological Food on Microbiota (CLEAR). Therefore, we will recruit 47 people to each group to have at least 40 at the end of the study. With 40 participants in each group, this analysis has >90% power to detect a 50% reduction in CO2e for the intervention group. To gain further insight into the development of intake of nutrients, CO2e, and the dietary sustainability score during the follow-up, we will use linear mixed models, with individual-specific baseline trajectories. Moreover, we will perform substitution analyses, i.e. scenarios where a number of meals high in CO2e are substituted for meals low in CO2e. Statistical analyses will be done in R-statistics.

ELIGIBILITY:
Inclusion Criteria:

- Preform office work ≤20 hours/week

Exclusion Criteria:

* Allergies excluding large food groups
* Visual or speech disability
* Not owning a smartphone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Change in dietary patterns and intake of fruit and vegetable | Baseline, after 4 weeks and after 8 weeks.
  Assessment of dietary patterns by the food-frequency questionnaire Meal-Q, expressed as servings per day or grams per day of meat, dairy products, fruit and vegetable.
Change from baseline in dietary carbon dioxide equivalents | Baseline, after 4 weeks and after 8 weeks.
  Assessment of dietary Carbon dioxide equivalents (CO₂e) by converting data from Meal-Q to a daily intake of 50 nutrients by linkage to the National Food Composition Table as well as to a database with Life cycle assessment (LCA) data for 65 different food products to calculate greenhouse gas emissions CO₂e per day.
Change in physical activity level | Baseline, after 4 weeks and after 8 weeks.
  Assessment of physical activity by the self-administrated Web-based questionnaire Active-Q, expressed as metabolic equivalent of task value (MET).
Changes in concentration of urinary pesticide residues in urine | Baseline, and after 8 weeks.
  Assessment of sustainable and organic food intake by measuring concentration of pesticide residues. Samples will be collected at two occasions; baseline (reference sample), and at the end (after 8 weeks) in 50ml FALCON polypropylene containers and stored at -80˚C until further analysis according to gold standard methods. The results will be calculated as μg pesticide/g creatinine to adjust for differences in urinary concentration.

SECONDARY OUTCOMES:
Changes in dietary sustainability score | Baseline, after 4 weeks and after 8 weeks
  Assessment of how the participants lifestyle correlate with the dietary sustainability score that we have developed. The score integrates measures of 14 factors related to lifestyle and sustainability, i.e. CO2e values.
Changes in the anthropometrical assessments (Body Mass Index) | Baseline, and after 8 weeks.
  Bodyweight (kg) and height (cm) measured using standardized procedures and equipment, including a stadiometer and bioelectrical impedance analysis. These measurements will be combined to calculate the Body Mass Index (BMI), which is reported in kg/m².
Stanford healthy Neighborhood Discovery Tool | Week 6, workshop number 5 of 6.
  An app that participants use to document factors that facilitate or hinder the participants from having a healthy or sustainable lifestyle to and from work and at work. The data consist of geo-coded photographs, text and audio narratives, and data on positive or negative attributes of the workplace (portrayed as a happy and sad smiley face in the app).
Experiences related to a healthy and sustainable lifestyle intervention | Week 8, workshop number 6 of 6.
  A web-based questionnaire that includes questions about what the participants think of the diet "likeability" that they have been assigned to and whether they may consider continuing eating according to the instructions after the study ends, and what potential obstacles they may have encountered.
Changes in intake of energy | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of energy in kilojoule/day (kJ/day) when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of energy in kJ by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of protein | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes changes in intake of protein in (g/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of protein in kJ by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of fat | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of fat in (kJ/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of fat in kJ by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of carbohydrates | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of carbohydrates in (kJ/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of macronutrients in kJ by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of dietary fiber | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of dietary fiber in (kJ/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of dietary fiber in kJ by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of vitamin A | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of vitamin A, measured in Retinol Equivalents per day (RE/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin A in RE by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of vitamin D | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of vitamin D, measured in micrograms per day (μg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin D in μg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of thiamin | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of thiamin, measured in milligrams per day (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of thiamin in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of riboflavin | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of riboflavin, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of riboflavin in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of niacin | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of niacin, measured in Niacin Equivalents per day (NE/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of niacin in NE by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of vitamin B6 | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of vitamin B6, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin B6 in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of folate | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of folate, measured in (μg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of folate in μg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of vitamin B12 | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of vitamin B12, measured in (μg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin B12 in μg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of vitamin C | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of vitamin C, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin C in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of calcium | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of vitamin C, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of vitamin C in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of phosphorus | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of phosphorus, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of phosphorus in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of potassium | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of potassium, measured in grams per day (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of potassium in g by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of iron | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of iron, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of iron in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of zinc | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of zinc, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of zinc in mg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of iodine | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of iodine, measured in (μg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of iodine in μg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in potassium | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of selenium, measured in (μg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of selenium in μg by linkage to the National Food Composition Table using the NutriCalc program.
Changes in intake of copper | Baseline, after 4 weeks and after 8 weeks.
  Assessment of changes in intake of copper, measured in (mg/day), when the participants shifts their diet from baseline to a healthy or sustainable lifestyle, using a validated food frequency questionnaire called Meal-Q. Questionnaire responses will be converted to daily intake of copper in mg by linkage to the National Food Composition Table using the NutriCalc program.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Bälter, PhD, Principal Investigator — Mälardalen University
Locations (1):
- Mälardalen University, Västerås, Västmanland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glympi A, Chasioti A, Balter K. Dietary Interventions to Promote Healthy Eating among Office Workers: A Literature Review. Nutrients. 2020 Dec 7;12(12):3754. doi: 10.3390/nu12123754. PMID 33297328
- [Background] Balter K. The importance of considering both nutrient quality and climate impact to support sustainable development. Am J Clin Nutr. 2021 Aug 2;114(2):412-413. doi: 10.1093/ajcn/nqab167. No abstract available. PMID 34091673
- See also: Official swedish project website — https://www.sofco.se/